CLINICAL TRIAL: NCT04737226
Title: The Association Between Ankle Mobility and Achilles Tendon, Plantar Fascia, Iliotibial Band Stiffness and Elasticity in Athletes
Brief Title: The Relation of Ankle Mobility and Achilles Tendon, Plantar Fascia and Iliotibial Band Mechanical Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Serkan Usgu, Assistant of professeur, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2020/100
Record Dates: First submitted 2021-01-20; First posted 2021-02-03 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Mobility Limitation; Stiffness of Right Ankle, Not Elsewhere Classified; Stiffness of Left Ankle, Not Elsewhere Classified; Tone Increased, Muscle
Keywords: Stiffness; Tone; Elasticity; Ankle mobility
MeSH Terms: conditions — Mobility Limitation; Muscle Hypertonia

STUDY DESIGN:
Intervention Model Description: Professional male athletes (basketballers, voleyballers, runners) will participate and divided to groups. AT, PF and ITB mechanical properties will evaluate with MyotonPro device (Myoton Ltd, Estonia). Ankle mobility will measure with inclinometer during a knee to wall lunge test.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Basketballers (Experimental)
  Interventions: Diagnostic Test: myotonometric assessment; Diagnostic Test: Ankle mobility assessment
- Volleyballers (Experimental)
  Interventions: Diagnostic Test: myotonometric assessment; Diagnostic Test: Ankle mobility assessment
- Runners (Experimental)
  Interventions: Diagnostic Test: myotonometric assessment; Diagnostic Test: Ankle mobility assessment

INTERVENTIONS:
Diagnostic Test: myotonometric assessment — The measurement method of the device is based on the free oscillation technique. Firstly, the probe of the device is placed perpendicular to the skin and a pre-pressure is applied to compress the subcutaneous tissue. Then, a short mechanical impulse is applied, causing damped oscillation on the tissue and the co-oscillation is recorded by an accelerometer.
Diagnostic Test: Ankle mobility assessment — The knee to wall lunge test will use in a standing position while the heel in contact with the ground and the knee was in line with second toe. Athletes will do lunge forward and inclinometer will be place at the middle anterior tibial crista and measurement will be record.

SUMMARY:
The myotonometric assessment is becoming popular and important in athletic population. It is mentioned an alternate method than expensive methods, and it is easy and reliable assessment. Still there is not enough information of mechanical characteristics in athletic population and ankle mobility. Most clinicians or trainers can use this results and technique for enhancing performance, rehabilitation or prevention

DETAILED DESCRIPTION:
The soft tissue mechanical properties can be assessed through elastography and ultrasonography. Both methods can measure passive and active soft tissue properties. These methods are the gold standard to measure stiffness and elasticity, but they are expensive, operator dependent and need a laboratory settings.Recently, myotonometric device has been used to measure the mechanical properties of the muscles and tendons. This method serves many advantages, such as non-invasive, painless and cost-effective. There is an increasing literature on athletic training about how training effects viscoelastic properties. However, to the best of our knowledge, there were no studies assessing stiffness and elasticity of AT, PF and ITB and the relation with ankle mobility in different sport disciplines. The purpose of this study were to demonstrate the mechanical properties of AT, PF and ITB and find out relation with restricted ankle mobility in athletes.

ELIGIBILITY:
Inclusion Criteria:

* being a professional athlete
* right dominant
* not having any lower extremity injury or surgery in the last 6 months,
* following routine training program.

Exclusion Criteria:

* a history of strain or surgery with knee or ankle,
* had any neurological or systemic disease.

Ages: 18 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Professional male athletes
Enrollment: 30 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Stiffness obtained from myotonometric assessment | through study completion, an average of 8 weeks
  Myoton device stimulations create natural oscillations in the tissue and records these oscillations using an accelerometer. Stiffness (N/m) is calculated by device.
Elasticity obtained from myotonometric assessment | through study completion, an average of 8 weeks
  Myoton device stimulations create natural oscillations in the tissue and records these oscillations using an accelerometer. Elasticity (log) is calculated by device.
Ankle range of motion | through study completion, an average of 8 weeks
  Inclinometer is be place at the middle anterior tibial crista during the knee to wall test. The angle of incliometer during a maximum distance between the largest toe and the wall that is recorded for ankle range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan kalyoncu üniversity, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cristi-Sanchez I, Danes-Daetz C, Neira A, Ferrada W, Yanez Diaz R, Silvestre Aguirre R. Patellar and Achilles Tendon Stiffness in Elite Soccer Players Assessed Using Myotonometric Measurements. Sports Health. 2019 Mar/Apr;11(2):157-162. doi: 10.1177/1941738118820517. Epub 2019 Jan 2. PMID 30601077
- [Background] Gavronski G, Veraksits A, Vasar E, Maaroos J. Evaluation of viscoelastic parameters of the skeletal muscles in junior triathletes. Physiol Meas. 2007 Jun;28(6):625-37. doi: 10.1088/0967-3334/28/6/002. Epub 2007 May 3. PMID 17664617
- [Background] Kubo K, Miyazaki D, Shimoju S, Tsunoda N. Relationship between elastic properties of tendon structures and performance in long distance runners. Eur J Appl Physiol. 2015 Aug;115(8):1725-33. doi: 10.1007/s00421-015-3156-2. Epub 2015 Mar 27. PMID 25813019
- [Background] Liu CL, Li YP, Wang XQ, Zhang ZJ. Quantifying the Stiffness of Achilles Tendon: Intra- and Inter-Operator Reliability and the Effect of Ankle Joint Motion. Med Sci Monit. 2018 Jul 14;24:4876-4881. doi: 10.12659/MSM.909531. PMID 30006997
- [Background] Pozarowszczyk B, Pawlaczyk W, Smoter M, Zarzycki A, Mroczek D, Kumorek M, Witkowski K, Adam K. Effects of Karate Fights on Achilles Tendon Stiffness Measured by Myotonometry. J Hum Kinet. 2017 Mar 12;56:93-97. doi: 10.1515/hukin-2017-0026. eCollection 2017 Feb. PMID 28469747